CLINICAL TRIAL: NCT05685342
Title: Comparison of the Opioid-sparing Effect of Preemptive and Preventive Intravenous Acetaminophen/Ibuprofen Fixed-dose Combination After Robot-assisted Radical Prostatectomy: A Double-blind Randomized Controlled Trial
Brief Title: Preemptive and Preventive Acetaminophen/Ibuprofen Fixed-dose Combination After Robot-assisted Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Kyongbo Pharmaceutical (Unknown)
Responsible Party: Principal Investigator, Hojin Lee, MD, PhD, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Maxigesic_Pre
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: A prospective randomized double-blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An investigator who is not involved in this study randomly allocates the group and another investigator who dose not evaluate clinical endpoints keeps the result of allocation in a sealed envelope.
  On the day of study, the second investigator opens the envelope to check allocation and sends a drug and normal saline in identical looking bottles with label only indicating the order of administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preemptive administration group (Experimental): Preemptive administration group will receive intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) for 15 minutes at the end of induction of anesthesia.
  Interventions: Drug: Acetaminophen/Ibuprofen fixed-dose combination
- Preventive administration group (Active Comparator): The preventive administration group will receive intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) for 15 minutes when surgical site closure starts.
  Interventions: Drug: Acetaminophen/Ibuprofen fixed-dose combination

INTERVENTIONS:
Drug: Acetaminophen/Ibuprofen fixed-dose combination — Intravenous administration of Acetaminophen (1000 mg)/Ibuprofen (300 mg) fixed-dose combination (total 100 ml)
  Other Names: Maxigesic

SUMMARY:
This prospective, randomized, double-blinded study is designed to compare opioid-sparing effect of preemptive and preventive intravenous acetaminophen/ibuprofen fixed-dose combination in patients undergoing robot-assisted radical prostatectomy (RARP). We hypothesize that preemptive administration of intravenous acetaminophen/ibuprofen fixed-dose combination can significantly reduce postoperative opioid consumption and pain severity than preventive administration in patients undergoing RARP.

DETAILED DESCRIPTION:
Adult patients undergoing elective robot-assisted radical prostatectomy are randomly allocated to receive preemptive administration of acetaminophen (1000 mg)/ibuprofen (300 mg) fixed-dose combination (n=77) or preventive administration (n=77). The preemptive administration group will receive intravenous acetaminophen (1000 mg)/ibuprofen (300 mg) for 15 minutes at the end of induction of anesthesia. The preventive administration group will receive same dosage of drug for same duration when surgical site closure starts.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective robot-assisted radical prostatectomy under general anesthesia
* American Society of Anesthesiologists (ASA) physical classification I-II
* Consent to IV-patient controlled analgesia use
* Willingness and ability to sign an informed consent document

Exclusion Criteria:

* Who do not understand or agree with our study
* American Society of Anesthesiologists (ASA) physical classification III-IV
* Chronic usage of opioid analgesics
* Moderate to severe pain with other cause before surgery
* Allergies to anesthetic or analgesic medications used in this study
* Anticipated blood loss larger than 2 liters
* Need for intensive care after surgery
* History of gastric ulcer or gastrointestinal bleeding
* History of liver failure, renal failure or heart failure
* Current alcoholism
* Taking anti-coagulation drugs or history of coagulation disease
* History of bronchial asthma
* Medical or psychological disease that can affect the treatment response
* Taking barbitutate or tricyclic antidepressant

Ages: 19 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Total fentanyl consumption during 24 hours | Postoperative 24 hours
  Postoperative fentanyl consumption (mcg) via IV patient controlled analgesia

SECONDARY OUTCOMES:
Total fentanyl consumption | Postoperative 2, 6, 48 hours
  Postoperative fentanyl consumption (mcg) via IV patient controlled analgesia (PCA)
Postoperative pain score | Postoperative 2 (resting only), 6, 24, 48 hours
  11-pointed NRS pain score at resting/coughing NRS (0-10): 0,"no pain"; 10, "worst pain imaginable"
Count of rescue analgesics administration | Postoperative 0-2, 2-6, 6-24, 24-48 hours
  Number of count of rescue analgesics administered because of patient's request for additional analgesia than IV PCA
Opioid side effects | Postoperative 0-2, 2-6, 6-24, 24-48 hours
  Incidence of opioid side effects like postoperative nausea/vomiting, hypotension, dizziness, somnolence and respiratory depression (%)
Quality of recovery-15 | Postoperative 24 hours
  Korean version of Quality of recovery-15 questionnaire (0-150): 0, "very poor recovery"; 150, "excellent recovery"

CONTACTS AND LOCATIONS:
Overall Officials: Hojin Lee, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided